CLINICAL TRIAL: NCT01565109
Title: Phase II Multicenter Study in the Preoperative Treatment of Gastric Adenocarcinoma Consisting of Chemotherapy Using Docetaxel-cisplatin-5FU + Lenograstim Followed by Chemoradiation Based 5FU and Oxaliplatin
Brief Title: NESC: Neoadjuvant Treatment of Gastric Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Recherche clinique (Other)
Responsible Party: Sponsor-Investigator, Recherche clinique, Doctor Laurent Mineur, Institut Sainte Catherine
Organization: Institut Sainte Catherine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NESC
Record Dates: First submitted 2010-10-13; First posted 2012-03-28 (Estimated); Last update posted 2025-01-22 (Actual); Status verified 2023-06

CONDITIONS: Gastric Adenocarcinoma
Keywords: NESC; NEOADJUVANT; GASTRIC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- Single arm study (Experimental): Docetaxel - Cisplatine - 5FU 2 cycles of Docetaxel - Cisplatine - 5 FU
  Radiation: Radiation of 45 Grays on 5 weeks Radiochemotherapy with Oxaliplatine (J1, J15 et J29) - 5FU on 5 weeks
  Interventions: Drug: Docetaxel - Cisplatine - 5FU; Radiation: Radiation of 45 Grays on 5 weeks

INTERVENTIONS:
Drug: Docetaxel - Cisplatine - 5FU — 2 cycles of Docetaxel - Cisplatine - 5 FU
Radiation: Radiation of 45 Grays on 5 weeks — Radiochemotherapy with Oxaliplatine (J1, J15 et J29) - 5FU on 5 weeks

SUMMARY:
It is estimated to 7300 the number of new cases of gastric cancer each year in France.

According to a randomized trial comparing 3 cycles of ECF (epirubicin, cisplatin, 5FU) administered before surgery and 3 cycles after surgery with surgery alone in adenocarcinoma of the stomach and lower esophagus, clinical and experimental data are the neoadjuvant chemotherapy is a new standard treatment for operable gastric cancer. This treatment with a median survival of more than 3 years to obtain a hazard ratio of 0.75 in favor of chemotherapy arm (p = 0.009). The 5-year survival being 36% for patients treated with chemotherapy versus 23% for surgery alone. Progression-free survival was also significantly prolonged with a hazard ratio of 0.66.

The proposed clinical study by Ajani et al shows that the combination of Docetaxel with the schema Cisplatin - 5FU provides greater clinical benefit and induces to consider the triple combination as a reference treatment in metastatic gastric cancer in patients under 65 years.

Preoperative radiochemotherapy is expected to increase the rate of curative resections, reduce gastrointestinal and hematologic toxicity.

Two studies evaluating the feasibility of preoperative RTCT in operable gastric adenocarcinoma with continuous 5GU (+ or - paclitaxel) and 45 Gy are available and the combination 5FU oxaliplatin has been assessed in the esophagus and rectum tumors.

The NESC study, Phase II, proposes the following schema: 2 cycles of chemotherapy with Docetaxel - Cisplatin - 5FU then preoperative chemoradiation with oxaliplatin - continuous 5FU and radiotherapy in locally advanced gastric adenocarcinoma stage III and IV non-metastatic administered before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, Age: 18 to 65
* ECOG performance status of ≤ 1
* Histological documentation of the gastric adenocarcinoma. An extension will be admitted to the omentum
* Adenocarcinoma of the stomach according to staging classification TNM Scannographic: T2bN0, T2bN1, T3NO T3N +, T4N0, and T4N + M0 (cardia, Siewert II, III, fundus, body, antrum) performed by ultrasonography and CT Scan. Optional : laparoscopy
* A positive peritoneal cytology is not a disqualifying factor if there is no macroscopic carcinomatosis
* Absence of previous abdominal irradiation above the 5th sacral vertebra (in the liver, pancreas, spleen, or mediastinal lodge)
* Loss of weight less than 15% over the base weight before diagnosis
* No psychological, familial, sociological or geographical condition that may affect compliance and adherence to treatment, patient monitoring or understanding of the study.
* Signed informed consent obtained before any study specific procedures.
* Food Consumption> 1000 calories / day whatever the mode of administration (enteral or parenteral)
* Laboratory test conducted within one week of starting to study treatment:

  * Absolute neutrophil count > 1500/mm3
  * Platelet count > 100 000/mm3
  * Total bilirubin <2 mg/dL
  * Serum creatinine <13 mg/dL or creatinine clearance > 40 ml/min
  * Hemoglobin (Hgb) ≥ 10 g/dL (Hemoglobin transfusion if necessary)
  * ALT / AST <1.5 x ULN
  * PTT ≥ 60 %
  * Life expectancy of at least 3 months

Exclusion Criteria:

* Peripheral sensory neuropathy ≥ grade 1 (according to CTCAE version 3.0).
* Myocardial infarction, stroke or pulmonary embolism, unstable angina less than 6 months before start of study drug.
* Uncontrolled infection
* Pregnant or breast-feeding patients. Women of childbearing potential must have a pregnancy test performed.
* Prior treatment for gastric adenocarcinoma
* Lower limbs arteritis (≥ stage II according the Leriche and Fontain classification)
* Patient participating in another clinical trial or already receiving other anti-cancer treatment
* Concomitant treatment with a phenytoin
* Known previous / current malignancy within the last 5 years except for non-melanoma skin, non-metastatic prostate carcinoma and cervival carcinoma in situ or superficial bladder carcinoma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Histological response rate on surgical specimen after chemotherapy and chemoradiotherapy preoperative | 1year
  Histological response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Sainte Catherine, Avignon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mineur L, Plat F, Desseigne F, Deplanque G, Belkacemi M, Moureau-Zabotto L, Beyrne CD, Jalali K, Obled S, Smith D, Vazquez L, Boustany R. NESC Multicenter Phase II Trial in the Preoperative Treatment of Gastric Adenocarcinoma with Chemotherapy (Docetaxel-Cisplatin-5FU+Lenograstim) Followed by Chemoradiation Based 5FU and Oxaliplatin and Surgery. Cancer Res Treat. 2024 Apr;56(2):580-589. doi: 10.4143/crt.2023.812. Epub 2023 Oct 5. PMID 37817565